CLINICAL TRIAL: NCT03959657
Title: Análisis de Una población en Edad Extrema de la Vida Con Fractura de fémur (Analysis of a Population in Extreme Age of Life With a Hip Fracture)
Brief Title: Analysis of a Population in Extreme Age of Life With a Hip Fracture
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-FEM-2017-17
Record Dates: First submitted 2018-10-25; First posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention performed by authors — Observational and retrospective study, no intervention performed

SUMMARY:
Observational retrospective study of pacients over 95 years admitted in traumatology ward with a osteoporotic hip fracture

ELIGIBILITY:
Inclusion Criteria:

* osteoporotic hip fracture

Exclusion Criteria:

Ages: 95 Years to 120 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients over 95 years
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days
Mortality | 3 months
Mortality | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Montserrat Barceló, Barcelona, Spain